CLINICAL TRIAL: NCT05194046
Title: A Randomized, Open-label, Multiple-dose, 3-way Crossover Phase 1 Clinical Trial to Evaluate Drug-drug Interactions and Safety Among JP-1366, Amoxicillin, and Clarithromycin in Healthy Volunteers
Brief Title: Drug-drug Interactions and Safety Among JP-1366, Amoxicillin, and Clarithromycin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: JP-1366-102
Record Dates: First submitted 2021-11-30; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Helicobacter Pylori Associated Gastrointestinal Disease
MeSH Terms: interventions — Amoxicillin; Capsules; Clarithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence A (Experimental): T1→Washout period(D6~14)→ T3→Washout period(D20~28)→ T2
  * T1: JP-1366 1capsule, 2 times per 1 day, repetition administration for 5 days
  * T2: amoxicillin 500mg 2 capsules + clarithromycin 500mg 1 tablet, 2 times per 1 day, repetition administration for 5 days
  * T3: JP-1366 1 capsule + amoxicillin 500mg 2 capsules + clarithromycin 500mg 1 tablet, 2 times per 1 day, repetition administration for 5 days
  Interventions: Drug: JP-1366 20mg 1capsule; Drug: Amoxicillin 500Mg Cap; Drug: Clarithromycin 500Mg Tab
- Sequence B (Experimental): T1 →Washout period(D6~14)→ T2→Washout period(D20~28) → T3
  * T1: JP-1366 1 capsule, 2 times per 1 day, repetition administration for 5 days
  * T2: amoxicillin 500mg 2 capsules + clarithromycin 500mg 1 tablet, 2 times per 1 day, repetition administration for 5 days
  * T3: JP-1366 1 capsule + amoxicillin 500mg 2 capsules + clarithromycin 500mg 1 tablet, 2 times per 1 day, repetition administration for 5 days
  Interventions: Drug: JP-1366 20mg 1capsule; Drug: Amoxicillin 500Mg Cap; Drug: Clarithromycin 500Mg Tab
- Sequence C (Experimental): T2 →Washout period(D6~14)→ T3→Washout period(D20~28) → T1
  * T1: JP-1366 1capsule, 2 times per 1 day, repetition administration for 5 days
  * T2: amoxicillin 500mg 2 capsules + clarithromycin 500mg 1 tablet, 2 times per 1 day, repetition administration for 5 days
  * T3: JP-1366 1 capsule + amoxicillin 500mg 2 capsules + clarithromycin 500mg 1 tablet, 2 times per 1 day, repetition administration for 5 days
  Interventions: Drug: JP-1366 20mg 1capsule; Drug: Amoxicillin 500Mg Cap; Drug: Clarithromycin 500Mg Tab
- Sequence D (Experimental): T2 →Washout period(D6~14)→ T1→Washout period(D20~28) → T3
  * T1: JP-1366 1 capsule, 2 times per 1 day, repetition administration for 5 days
  * T2: amoxicillin 500mg 2 capsules + clarithromycin 500mg 1 tablet, 2 times per 1 day, repetition administration for 5 days
  * T3: JP-1366 1 capsule + amoxicillin 500mg 2 capsules + clarithromycin 500mg 1 tablet, 2 times per 1 day, repetition administration for 5 days
  Interventions: Drug: JP-1366 20mg 1capsule; Drug: Amoxicillin 500Mg Cap; Drug: Clarithromycin 500Mg Tab
- Sequence E (Experimental): T3 →Washout period(D6~14)→ T1→Washout period(D20~28) → T2
  * T1: JP-1366 1 capsule, 2 times per 1 day, repetition administration for 5 days
  * T2: amoxicillin 500mg 2 capsules + clarithromycin 500mg 1 tablet, 2 times per 1 day, repetition administration for 5 days
  * T3: JP-1366 1 capsule + amoxicillin 500mg 2 capsules + clarithromycin 500mg 1 tablet, 2 times per 1 day, repetition administration for 5 days
  Interventions: Drug: JP-1366 20mg 1capsule; Drug: Amoxicillin 500Mg Cap; Drug: Clarithromycin 500Mg Tab
- Sequence F (Experimental): T3 →Washout period(D6~14)→ T2→Washout period(D20~28) → T1
  * T1: JP-1366 1 capsule, 2 times per 1 day, repetition administration for 5 days
  * T2: amoxicillin 500mg 2 capsules + clarithromycin 500mg 1 tablet, 2 times per 1 day, repetition administration for 5 days
  * T3: JP-1366 1 capsule + amoxicillin 500mg 2 capsules + clarithromycin 500mg 1 tablet, 2 times per 1 day, repetition administration for 5 days
  Interventions: Drug: JP-1366 20mg 1capsule; Drug: Amoxicillin 500Mg Cap; Drug: Clarithromycin 500Mg Tab

INTERVENTIONS:
Drug: JP-1366 20mg 1capsule — will be orally administered
Drug: Amoxicillin 500Mg Cap — Amoxicilin 500Mg 2 capsules will be orally administered
Drug: Clarithromycin 500Mg Tab — Amoxicilin 500Mg 1 tablet will be orally administered

SUMMARY:
To evaluate the effect of coadministration of amoxicillin and clarithromycin on safety, tolerability and pharmacokinetics of JP-1366 in healthy subjects and the effect of JP-1366 on safety, tolerability and pharmacokinetics of amoxicillin and clarithromycin in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Subject who has fully informed about this study and understand completely, decide to participate voluntarily and agree with the written consent approved by the IRB in Bundang Cha hospital before screening test.
* A healthy volunteer in the age of upper 19 at the time of the screening test.
* Subject whose BMI was 18.0 or more and 30.0 or less and whose body weight was 50kg or more if in male, and 45kg or more if in female at the same time.

  * Body Mass Index (BMI) = Body weight(kg) / Height(m)2

Exclusion Criteria:

1. Medical History

1. The Subject who has clinically significant diseases with liver, kidney, nervous system, digestive system, respiratory system, and endocrine system, musculoskeletal system or the blood or tumor disease, cardiovascular disease (including orthostatic hypotension), mental disorder or with history of the disease.
2. The subject who has a history of gastrointestinal disorders (gastrointestinal ulcers, gastritis, gastric ulcer, gastroesophageal reflux disease, Crohn's disease, etc.) or history of gastrointestinal surgery that may affect the safety and PK/PD Evaluation of the investigational product (Except for simple cecal surgery and hernia surgery)
3. The subject who has a hereditary disorder (galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption etc.).

2. Allergy drug hypersensitivity and drug abuse

1. The subject with clinically significant hypersensitivity reactions (Except a slight allergic rhinitis which is no need to administration).
2. The subject with the history of hypersensitivity reactions to the investigational product, the ingredients in investigational product (FCF, Sunset Yellow FCF), Digestive ulcer drugs and other drugs (aspirin, antibiotics, etc.)
3. The subject who has a history of drug abuse or who has tested positive for an abuse drug in a drug screening test.

3. Laboratory Test

1. Vital Sign Measures of resting blood pressure while the subject remained in the sitting position for at least 3 minutes. Systolic > 150 mmHg or < 90 mmHg, or diastolic > 100 mmHg or < 50 mmHg.
2. Screening laboratory test showing any of the following abnormal laboratory results:

   - ALT, AST, Total bilirubin > 2.0 x ULN
   * e-GFR < 60 mL/min/1.73m2 (CKD-EPI formula)
   * Positive result for Serological test (HBsAg, HCV Ab, HIV Ab, Syphilis regain test)
3. Clinically significant ECG abnormalities

4. Prohibited medication and therapy

1. The subject taking drug of enzyme induction or inhibition within one month prior to the first scheduled drug administration.
2. The subject who has participated in other clinical trials or bioequivalence studied and received and received clinical trial drug or bioequivalence study drug, within 6 months prior to the first scheduled drug administration.
3. The subject taking any prohibited drug or herbal medicine, OTC drugs or vitamin within 2 weeks prior to the first scheduled drug administration.
4. The subject who has taken any diet which affect to drug metabolism (Grapefruit juice, Broccoli, Garlic extract etc.) within 3 days prior to the first scheduled drug administration or who cannot be forbidden the ingestion of it.

5. Donating and Receiving blood

1. The subject who did a whole blood donation within 2 months prior to the first scheduled drug administration or a component blood donation (pheresis) within one month
2. The subject who has received blood transfusions within one month prior to the first scheduled drug administration.

6. Pregnant and Contraception

1. Pregnant and Lactating women
2. Subjects who do not agree to use medically acceptable methods of contraception during the period study - Use of an intrauterine device - Use of barrier contraception (for men or women) and using spermicidal at the same time - Vasectomy, tubectomy, tubal ligation, hysterectomy

7. And others

1. Subjects who are judged unsuitable to participate in the study in the opinion of the investigator
2. The subject who continue to drink (over 21units/week, 1 unit = 10g of pure alcohol) within 6 months from screening or who cannot abstain from drinking during the clinical trial period from 3days before the first administration date.
3. The subject whose average smoking amount exceeds 10 cigarettes per day within 6 months.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Cmax,ss of JP-1366, Amoxicillin, Clarithromycin | The time of steady state (after repetition administration for 5 days)
AUCτ of JP-1366, Amoxicillin, Clarithromycin | The time of steady state (after repetition administration for 5 days)

SECONDARY OUTCOMES:
Tmax of JP-1366, Amoxicillin, Clarithromycin, 14-OH-Clarithromycin | The time of steady state (after repetition administration for 5 days)
t1/2 of JP-1366, Amoxicillin, Clarithromycin, 14-OH-Clarithromycin | The time of steady state (after repetition administration for 5 days)
CLss/F of JP-1366, Amoxicillin, Clarithromycin, 14-OH-Clarithromycin | The time of steady state (after repetition administration for 5 days)
Vdss/F of JP-1366, Amoxicillin, Clarithromycin, 14-OH-Clarithromycin | The time of steady state (after repetition administration for 5 days)
Cmax,ss of 14-OH-Clarithromycin | The time of steady state (after repetition administration for 5 days)
AUCτ of 14-OH-Clarithromycin | The time of steady state (after repetition administration for 5 days)
14-OH-Clarithromycin/Clarithromycin metabolic ratio | The time of steady state (after repetition administration for 5 days)

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Through study completion, an average of 46 days
  Vital sign, Physical examination, Laboratory test, 12-lead ECG, Prior/ Concomitant medication, Adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- Cha University Bundang Medical Center, Gyeonggi-do, South Korea